CLINICAL TRIAL: NCT03004001
Title: Effect of PCSK9-Antibody (Alirocumab) on Dyslipidemia Secondary to Nephrotic Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Difficult recruitment
Sponsor: Gloria Vega (U.S. Federal Agency)
Collaborators: Regeneron Pharmaceuticals (Industry); Aventis Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Gloria Vega, Principal Investigator at Dallas VA Medical Center, Dallas VA Medical Center
Organization: Dallas VA Medical Center (U.S. Federal Agency)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: VA16-029
Record Dates: First submitted 2016-12-16; First posted 2016-12-28 (Estimated); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Nephrotic Syndrome
Keywords: Severe proteinuria; Dyslipidemia
MeSH Terms: conditions — Nephrotic Syndrome; Proteinuria; Dyslipidemias | interventions — alirocumab; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alirocumab and atorvastatin (Experimental): Alirocumab 150 mg bi-weekly and atorvastatin 20 mg/d
  Interventions: Drug: Alirocumab; Drug: Atorvastatin
- Alirocumab placebo and atorvastatin (Placebo Comparator): Alirocumab placebo biweekly and atorvastatin 20 mg/d
  Interventions: Drug: Alirocumab placebo; Drug: Atorvastatin

INTERVENTIONS:
Drug: Alirocumab — 150 mg biweekly
  Other Names: Praluent
  Arms: Alirocumab and atorvastatin
Drug: Alirocumab placebo — placebo
  Other Names: Praluent placebo
  Arms: Alirocumab placebo and atorvastatin
Drug: Atorvastatin — 20 mg/day
  Other Names: Lipitor

SUMMARY:
The study purpose is to determine the hypolipidemic effect of Alirocumab co-administered with atorvastatin on levels of triglyceride-rich lipoproteins and LDL compared to monotherapy with atorvastatin in patients with dyslipidemia secondary to nephrotic syndrome.

DETAILED DESCRIPTION:
The trial is randomized (1:1 alirocumab to placebo), double-blinded, placebo-controlled with a cross-over design. The trial will last 10 months and includes a 10 week washout period between study phases.Twenty adult subjects with dyslipidemia secondary to nephrotic syndrome and treated with atorvastatin will be recruited. Alirocumab or placebo will be co-administered biweekly. Safety, efficacy chemistries, vital signs, anthropometry and monitoring for adverse events also will done at each visit.

ELIGIBILITY:
Inclusion Criteria:

* Nephrotic Syndrome (NS) (FSGS, IMN or NS and type 2 DM)
* atorvastatin
* LDL C >= 70 mg/dl or non-HDL C >= 100 mg/dl
* Plasma trigycerides < 800 mg/dl.
* Highly effective methods of contraception for pre-menopausal women
* Post-menopausal women must be amenorrheic for at least 12 months.

Exclusion Criteria:

* homozygous FH
* Fibrates within 6 weeks of screening visit
* Uncontrolled hypothyroidism
* Known history of hemorrhagic stroke
* Known history of loss of function of PCSK9
* use of systemic corticosteroids unless used as replacement therapy for pituitary/adrenal disease with a stable regimen for at least 6 weeks of randomization
* Previous treatment with at least a single dose of alirocumab or any other anti-PCSK9 monoclonal antibody
* Other conditions or situations per protocol
* Laboratory findings or contraindications to background therapies
* Warnings/precautions of use (when appropriate) as displayed in the respective national product labeling
* Any currently known contra-indication to study drug, pregnancy or breastfeeding of infants.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2017-01; Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Levels of plasma lipoproteins | up to 10 months
  ion mobility lipoprotein analysis

SECONDARY OUTCOMES:
Levels of PCSK9 | up to 10 months
  immunoassay
Triglyceride-rich lipoproteins (Remnants) | up to 10 months
  immunoassay
Lipidomics | up to 10 months
  mass spectroscopy

CONTACTS AND LOCATIONS:
Overall Officials: Gloria L Vega, PhD, Principal Investigator — Dallas VAMC; Yin Oo, MD, Study Director — Dallas VA Medical Center; Michael Concepcion, MD, Study Director — Dallas VA Medical Center
Locations (1):
- DallasVAMC, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Vega GL, Grundy SM. Lovastatin therapy in nephrotic hyperlipidemia: effects on lipoprotein metabolism. Kidney Int. 1988 Jun;33(6):1160-8. doi: 10.1038/ki.1988.125. PMID 3165483
- [Background] Toto RD, Grundy SM, Vega GL. Pravastatin treatment of very low density, intermediate density and low density lipoproteins in hypercholesterolemia and combined hyperlipidemia secondary to the nephrotic syndrome. Am J Nephrol. 2000 Jan-Feb;20(1):12-7. doi: 10.1159/000013549. PMID 10644862
- [Background] Vega GL, Toto RD, Grundy SM. Metabolism of low density lipoproteins in nephrotic dyslipidemia: comparison of hypercholesterolemia alone and combined hyperlipidemia. Kidney Int. 1995 Feb;47(2):579-86. doi: 10.1038/ki.1995.73. PMID 7723244
- [Background] Jin K, Park BS, Kim YW, Vaziri ND. Plasma PCSK9 in nephrotic syndrome and in peritoneal dialysis: a cross-sectional study. Am J Kidney Dis. 2014 Apr;63(4):584-9. doi: 10.1053/j.ajkd.2013.10.042. Epub 2013 Dec 4. PMID 24315769